CLINICAL TRIAL: NCT01609946
Title: Evaluation of Realtime-Elastography for Differentiation of Thyroid Nodules: a Multicenter Study
Brief Title: Realtime-Elastography (RTE) and Thyroid Nodules
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Vermehren (Other)
Responsible Party: Sponsor-Investigator, Johannes Vermehren, Record Keeper, Johann Wolfgang Goethe University Hospital
Organization: Johann Wolfgang Goethe University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: JWGUHMED1-004
Record Dates: First submitted 2012-05-30; First posted 2012-06-01 (Estimated); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Thyroid Nodules
Keywords: presenting for FNAB or surgery
MeSH Terms: conditions — Thyroid Nodule | interventions — Cytological Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Realtime-Elastography, linear ultrasound probe, Hitachi EUB-900, Japan
Procedure: Cytology (FNAB) or Surgery

SUMMARY:
The study is an open, prospective multicenter study. According to the statistical sample size calculation 593 patients with thyroid nodules ≥ 5mm in size will be included in the study. Reference methods are cytology obtained by Fine needle aspiration biopsy (FNAB) or histology obtained by surgery.

All patients will receive an B-mode and Duplex ultrasound examination of the thyroid gland, as well as Realtime Elastography of thyroid nodules.

Results of B-mode and Duplex ultrasound are compared to Realtime Elastography to evaluate the additional value of Realtime Elastography in the diagnostic work up of thyroid nodules.

ELIGIBILITY:
Inclusion Criteria:

* patients with thyroid nodules ≥ 5mm in size and TSH ≥ 0,35µU/ml
* Cytology obtained by FNAB or thyroid surgery planned
* age ≥ 18 year
* signed written consent

Exclusion Criteria:

* Diseases which preclude study accomplishment or put the patient at any risk (e.g. psychiatric diseases)
* Non-contractually capable persons
* Pregnancy
* Lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 602 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Realtime-Elastography scores I-IV in thyroid nodules
  Scores: I-II: benign; III-IV: malignant nodules. The sensitivity and specificity of Realtime-Elastography for the diagnosis of malignant thyroid nodules will be calculated on the basis of above-specified criteria. Cytology is used as reference method for benign nodules and histology for malignant nodules.

SECONDARY OUTCOMES:
Comparison of Realtime-Elastography with B-mode and Duplex-Ultrasonography concerning the additional diagnostic information obtained by Realtime-Elastography

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Bojunga, MD, Principal Investigator — Klinikum der J. W. Goethe-Universität, Frankfurt, Germany
Locations (10):
- Germany (10):
  - Caritas-Krankenhaus, Bad Mergentheim
  - Klinikum Bielefeld, Bielefeld
  - Bürgerhospital, Frankfurt
  - Klinikum der J. W. Goethe-Universität, Frankfurt am Main
  - Helfenstein Klinik, Geislingen
  - Universitätsklinikum Leipzig, Leipzig
  - Klinikum am Steinberg, Reutlingen
  - Endokrinologie und Diabetologie im Zentrum, Stuttgart
  - Universitätsklinikum Ulm, Ulm
  - Deutsche Klinik für Diagnostik, Wiesbaden